CLINICAL TRIAL: NCT01801709
Title: A Phase I/II, Open Labeled, Monocentric Study of Direct Intracranial Administration of a Replication Deficient Adeno-associated Virus Gene Transfer Vector Serotype rh.10 Expressing the Human ARSA cDNA to Children With Metachromatic Leukodystrophy.
Brief Title: Intracerebral Gene Therapy for Children With Early Onset Forms of Metachromatic Leukodystrophy
Acronym: TG-MLD
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Collaborators: European Leukodystrophy Association (Other); Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C11-09; 2011-004410-42 (EudraCT Number)
Record Dates: First submitted 2013-01-28; First posted 2013-03-01 (Estimated); Last update posted 2025-11-18 (Actual); Status verified 2025-01

CONDITIONS: Metachromatic Leukodystrophy
Keywords: Brain Gene Therapy; Adeno Associated vector; Lysosomal sotage diseases; Leukodystrophies
MeSH Terms: conditions — Leukodystrophy, Metachromatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- AAVrh.10cuARSA (Experimental): intracerebral administration of AAVrh.10cuARSA at 12 sites in the white matter of both brain hemispheres.
  Interventions: Genetic: intracerebral administration of AAVrh.10cuARSA

INTERVENTIONS:
Genetic: intracerebral administration of AAVrh.10cuARSA

SUMMARY:
The objective of this open-label, single arm, monocentric, phase I/II clinical study is to assess safety and efficacy of ARSA gene transfer in the brain of children affected with early onset forms of Metachromatic Leukodystrophy (MLD). For this purpose, an adeno-associated virus serotype rh.10 (AAVrh.10) vector will be used to transfer the ARSA cDNA coding for Arylsulfatase A (ARSA) enzyme into the brain of children. Five patients with early onset form of MLD, age ranging from 6 months to 4 years, will be included in this protocol and will be followed during 24 months.

Patients will be selected at presymptomatic or early stage of their disease, following clinical, neuropsychological and brain imaging criteria.

Twelve simultaneous injections of the investigational medicinal product will be performed in the white matter of both brain hemispheres, through 6 image-guided tracks, with 2 deposits per track.

A low dose (1x10EXP12 vg total) will be administered to the first 2 patients, while the last 3 will receive a higher dose (4x10EXP12 vg total).

Safety and efficiency will be evaluated based on clinical, neuropsychological, radiological, electrophysiological and biological parameters.

ELIGIBILITY:
Inclusion Criteria:

* Boys or girls with an early onset form of MLD.
* Age between 6 months and 5 years, inclusive
* Diagnostic of MLD based on the measurement of ARSA activity in leukocytes and the accumulation of sulfatides in urine, along with normal activity of at least one other sulfatase
* Informed consent signed up and willingness for monitoring 2 years after treatment.
* Normal values for standard laboratory tests

Exclusion Criteria:

* Absence of ARSA protein by immunocytochemistry and/or ELISA
* Gestational age <32 weeks of amenorrhoea and age < 1 year
* Brain atrophy with a subdural space > 10 mm in the frontal region
* Performance IQ<50 at WPPSI-III or cognitive function < 3rd percentile at the Bayley's test of infant development
* If age > 16 months at inclusion, inability to walk few steps alone OR inability to walk few steps with support on one side along with inability to stand up alone
* Impossibility for anesthesia
* Malignancy, cardiac malformation, liver dysfunction, or renal dysfunction
* Neurological disorder, except benign, not related to MLD.
* Any other clinically significant untreated co-morbid medical condition as determined by the clinical investigator, including cardiac, pulmonary or kidney disease.
* MRI impossibility
* Evoked potential impossibility
* Participation to another therapeutic clinical trial for MLD.
* Unaffiliated to any French or any other National Health Insurance.

Ages: 6 Months to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 5 (Actual)
Dates: Start 2014-06 (Actual); Primary Completion 2016-06 (Actual); Study Completion 2022-12-20 (Actual)

PRIMARY OUTCOMES:
Evaluate the tolerance of the intracerebral administration of a single dose of AAVrh.10cuARSA | During the two years follow-up
  Tolerance will be measured by :
  * Adverse event,
  * Clinical and neurological exams,
  * Laboratory tests,
  * Neuroimagery (CT scan, brain MRI).

SECONDARY OUTCOMES:
Evaluate the efficacy of intracerebral administration of a single dose of AAVrh.10cuARSA to stop the disease progression. | During the two years follow-up
  Efficacy will be measured by:
  * MLD neurological severity score,
  * Neurological evaluation,
  * Motor scores (GMFM, Ashworth and ICARS),
  * Cognitive functions (Bayley Scales of Infant Development (BSID)(0-42 months), or Wechsler Preschool and Primary Scale of Intelligence-III (WPPSI-III) (43 months-6 years)),
  * MLD severity MRI score, MRI-DTI parameters, measurement of cerebral atrophy and spectroscopy,
  * Neuroelectrophysiological tests (peripheral nerve conduction velocity, visual, auditory and somatosensory evoked potentials).

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Aubourg, MD-PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris and Institut National de la Santé et de la Recherche Médicale; Caroline Sevin, MD-PhD, Study Director — Assistance Publique - Hôpitaux de Paris; Michel Zerah, MD, PhD, Study Director — Assistance Publique - Hôpitaux de Paris; Thomas Roujeau, MD, PhD, Study Director — Assistance Publique - Hôpitaux de Paris; Nathalie Cartier, MD, PhD, Study Director — Institut National de la Santé et de la Recherche Biomédicale
Locations (1):
- Bicêtre Hospital - Paris Sud, Le Kremlin-Bicêtre, France

REFERENCES:
- [Background] Piguet F, Sondhi D, Piraud M, Fouquet F, Hackett NR, Ahouansou O, Vanier MT, Bieche I, Aubourg P, Crystal RG, Cartier N, Sevin C. Correction of brain oligodendrocytes by AAVrh.10 intracerebral gene therapy in metachromatic leukodystrophy mice. Hum Gene Ther. 2012 Aug;23(8):903-14. doi: 10.1089/hum.2012.015. Epub 2012 Jul 23. PMID 22642214
- [Background] Sondhi D, Johnson L, Purpura K, Monette S, Souweidane MM, Kaplitt MG, Kosofsky B, Yohay K, Ballon D, Dyke J, Kaminksy SM, Hackett NR, Crystal RG. Long-term expression and safety of administration of AAVrh.10hCLN2 to the brain of rats and nonhuman primates for the treatment of late infantile neuronal ceroid lipofuscinosis. Hum Gene Ther Methods. 2012 Oct;23(5):324-35. doi: 10.1089/hgtb.2012.120. Epub 2012 Nov 6. PMID 23131032
- [Background] Colle MA, Piguet F, Bertrand L, Raoul S, Bieche I, Dubreil L, Sloothaak D, Bouquet C, Moullier P, Aubourg P, Cherel Y, Cartier N, Sevin C. Efficient intracerebral delivery of AAV5 vector encoding human ARSA in non-human primate. Hum Mol Genet. 2010 Jan 1;19(1):147-58. doi: 10.1093/hmg/ddp475. PMID 19837699
- [Background] i Dali C, Hanson LG, Barton NW, Fogh J, Nair N, Lund AM. Brain N-acetylaspartate levels correlate with motor function in metachromatic leukodystrophy. Neurology. 2010 Nov 23;75(21):1896-903. doi: 10.1212/WNL.0b013e3181feb217. PMID 21098404
- [Result] Zerah M, Piguet F, Colle MA, Raoul S, Deschamps JY, Deniaud J, Gautier B, Toulgoat F, Bieche I, Laurendeau I, Sondhi D, Souweidane MM, Cartier-Lacave N, Moullier P, Crystal RG, Roujeau T, Sevin C, Aubourg P. Intracerebral Gene Therapy Using AAVrh.10-hARSA Recombinant Vector to Treat Patients with Early-Onset Forms of Metachromatic Leukodystrophy: Preclinical Feasibility and Safety Assessments in Nonhuman Primates. Hum Gene Ther Clin Dev. 2015 Jun;26(2):113-24. doi: 10.1089/humc.2014.139. Epub 2015 Apr 28. PMID 25758611